CLINICAL TRIAL: NCT01906866
Title: A Randomized, Placebo-controlled Study to Investigate the Efficacy and Safety of Circadin® to Alleviate Sleep Disturbances in Children With Neurodevelopmental Disabilities
Brief Title: Efficacy and Safety of Circadin® in the Treatment of Sleep Disturbances in Children With Neurodevelopment Disabilities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU_CH_7911
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disorders
Keywords: Sleep disturbance; Circadian; Prolong release melatonin; Autism Spectrum Disorder; Smith-Magenis Syndrome; Angelman Syndrome; tuberous sclerosis
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias; Autism Spectrum Disorder; Smith-Magenis Syndrome; Angelman Syndrome; Tuberous Sclerosis | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circadin 2/5/10 mg (Active Comparator): Active arm
  Interventions: Drug: Circadin 2/5/10 mg
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Circadin 2/5/10 mg — Circadin 2/5/10 mg. Active arm
  Other Names: Active arm
  Arms: Circadin 2/5/10 mg
Drug: Placebo — Control arm
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the efficacy and safety of Circadin in children with neurodevelopmental disorders and to determine the dose, this randomized, placebo-controlled study is planned to evaluate the efficacy of a double-blind, 13 week treatment period with Circadin 2/5mg in improving maintenance of sleep, sleep latency and additional parameters in children with neurodevelopmental disabilities. The efficacy and safety of Circadin 2/5 mg will continue to be assessed during an open-label extension period of 13 weeks.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled study in children diagnosed with autism spectrum disorders (ASDs) and neurodevelopmental disabilities caused by neurogenetic diseases.

Children who are found to be eligible for the study will follow a 4-week, basic sleep hygiene and behavioral intervention wash-out period, and will continue in a 2-week single-blind (SB) placebo run-in period. Then, they will be randomized in a 1:1 ratio to receive either Circadin® 2 mg or placebo for 3 weeks in a double-blind treatment period.

After 3 weeks of treatment, on the last day of Week 5 ±3 days (Visit 3), sleep variables will be assessed to determine if dose modification (an increase to 5 mg) is required. Children will then continue on 2 or 5 mg of Circadin® or placebo for an additional double-blind period of 10 weeks. This double-blind period will be followed by an open-label period of 13 weeks. At the end of the 13-week open-label period on the last day of Week 28 ±3 days (Visit 5), sleep variables will be assessed to determine if a potential additional dose modification (i.e., an increase either to 5 mg for patients who are still on 2 mg or an increase to 10 mg for patients who are on 5 mg) is necessary (If a dose increase is decided upon, the dose increase should be from 2 mg to 5 mg, or 5 mg to 10 mg). Children will continue at 2, 5, or 10 mg Circadin® in an open-label period for another 78 weeks of follow-up, which will include continuous safety monitoring and 2 efficacy assessment time points at Weeks 41 and 54. The study will end with a 2-week SB placebo run-out period.

Each patient will participate in the study until the end of the second open-label safety follow-up period, and 2 week run-out period. The study duration will be 112 weeks, including the 4-week wash-out period with sleep hygiene and behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, all patients must satisfy all of the following criteria at screening:

1. Must be children 2 to 17.5 years of age at Visit 2 who comply with taking the study drug
2. Must have written informed consent provided by a legal guardian and assent (if needed)
3. Must have a documented history of ASD according to or consistent with the ICD-10 (International Classification of Diseases) or DSM-5/4 (Diagnostic and Statistical Manual of Mental Disorders) criteria, or neurodevelopmental disabilities caused by neurogenetic diseases (i.e., Smith-Magenis syndrome, Angelman syndrome, Bourneville's disease [tuberous sclerosis]) as confirmed by case note review showing that diagnosis was reached through assessment by a community pediatrician or pediatric neurologist or other health care professionals experienced in the diagnosis who took into account early developmental history and school records.
4. Must have current sleep problems including: a minimum of 3 months of impaired sleep defined as ≤6 hours of continuous sleep AND/OR ≥0.5 hour sleep latency from light off in 3 out of 5 nights based on parent reports and patient medical history. (The maintenance and latency problems do not necessarily have to be in the same 3 nights of the week.)
5. May be on a stable dose of non-excluded medication for 3 months, including anti- epileptics, anti-depressants (selective serotonin reuptake inhibitors [SSRIs]), stimulants, all mood changing drugs and β-blockers. (Only morning administration of β-blockers is allowed since β-blockers at night have the potential to reduce endogenous melatonin levels and might cause disturbed sleep)
6. The sleep disturbance is not due to the direct physiological effects of any concomitant medications such as SSRIs, stimulants, etc.

After completing 4 weeks of sleep hygiene training (for those who need it) and 2 weeks of placebo run-in, patients will be eligible to continue the study if they comply with the following:

* Continue to fulfill sleep problem criteria (see Inclusion Criterion 4) based on the completed Sleep and Nap Diary entered into the electronic case report form
* Parents demonstrate compliance in Sleep and Nap Diary completion (5 out of 7 nights). Compliance means that in at least 5 out of 7 nights per week (total of 2 weeks before each scheduled visit) the parents complete the diary pages with all mandatory questions
* Continue to fulfil all other eligibility criteria

Exclusion Criteria:

Children who meet any of the following criteria will be excluded from participating in the study:

1. Have had treatment with any form of melatonin within 2 weeks prior to Visit 1
2. Have a known allergy to melatonin or lactose
3. Have a known moderate to severe sleep apnea
4. Have an untreated medical/ineffectively treated/psychological condition that may be the etiology of sleep disturbances
5. Did not respond to previous Circadin® therapy based on past medical history records in the last 2 years
6. Are taking or have been taking prohibited medication within 2 weeks prior to Visit 1 (Section 7.1)
7. Are females of child-bearing potential that are not using contraceptives and/or breastfeeding and that are sexually active (Abstinence is an acceptable method of contraception.)
8. Pregnant females
9. Are currently participating in a clinical trial or have participated in a clinical trial involving medicinal product within the last 3 months prior to the study [this does not include patients who participated in the Phase I Pharmacokinetics (PK) study who can be already included in the study]
10. Children with known renal or hepatic insufficiency

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2013-10; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gringras, PhD, Principal Investigator — Thoma's Hospital, Westminster Bridge Rd, London; Robert Findling, MD, Principal Investigator — Kennedy Krieger Institute, Baltimore, Maryland, USA
Locations (28):
- United States (18):
  - Southwest Autism Research and Resource Center (SARRC), Phoenix, Arizona
  - Crystal BioMedical Research, LLC, Miami Lakes, Florida
  - Lake Mary Pediatrics, Orange City, Florida
  - Mate Lazlo, West Palm Beach, Florida
  - Attalla Consultants LLC, dba Institue for Behabiovral medicine, Smyrna, Georgia
  - AMR Baber research INC, Naperville, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Child Neurology Specialists/ CRCN, Henderson, Nevada
  - Clinical research center of New Jersey, LLC, Voorhees Township, New Jersey
  - Geinsinger Clinic, Danville, Pennsylvania
  - The children's hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - INSITE Clinical Research, DeSoto, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
  - Ericksen Research & Development, Clinton, Utah
  - Pacific institute of medical science, Bothell, Washington
- Helsinki Sleep Clinic Vitalmed OY, Helsinki, Finland
- France (2):
  - Hospital Raymond Poincare, Garches
  - Strasbourg University Hospital Depatment of Child Psychiatry & Neurology, Strasbourg
- Netherlands (3):
  - Yulius Mental Health Organization, Dordrecht
  - Hospital Gelderse Vallei, Ede
  - University Medical Center Groningen, Groningen
- United Kingdom (4):
  - Birmingham Childrens Hospital NHS FOUNDATION TRUST, Birmingham
  - Blackpool Victoria Teaching Hospitals NHS Foundation Trust, Blackpool
  - Guy's & St. Thomas's NHS Foundation Trust of St Thomas's Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Malow BA, Findling RL, Schroder CM, Maras A, Breddy J, Nir T, Zisapel N, Gringras P. Sleep, Growth, and Puberty After 2 Years of Prolonged-Release Melatonin in Children With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2021 Feb;60(2):252-261.e3. doi: 10.1016/j.jaac.2019.12.007. Epub 2020 Jan 23. PMID 31982581
- [Derived] Gringras P, Nir T, Breddy J, Frydman-Marom A, Findling RL. Efficacy and Safety of Pediatric Prolonged-Release Melatonin for Insomnia in Children With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2017 Nov;56(11):948-957.e4. doi: 10.1016/j.jaac.2017.09.414. Epub 2017 Sep 19. PMID 29096777

RESULTS

PARTICIPANT FLOW:
Groups:
- Circadin 2/5/10 mg: Circadin 2/5/10 mg: Active arm
- Placebo: Placebo arm
  Placebo
Period: Overall Study
Arm/Group | Circadin 2/5/10 mg | Placebo
Started | 60 | 65
Completed | 51 | 44
Not Completed | 9 | 21

BASELINE CHARACTERISTICS:
Population: All patients in the Safety Analysis Set who satisfied all major entry criteria (Criteria 1-5) and who had a valid mean TST result recorded for baseline and at least one post-baseline period assessment during the double blind phase. Patients were classified according to randomized treatment. This analysis set was used for all efficacy analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Circadin 2/5/10 mg | Placebo | Total
Number analyzed (Participants) | 60 | 65 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 65 | 125
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (4.08) | 8.4 (4.24) | 8.7 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 45 | 47 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 8 | 9
  White | 57 | 55 | 112
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 5 | 4 | 9
  United States | 44 | 50 | 91
  Finland | 0 | 1 | 1
  United Kingdom | 8 | 8 | 16
  France | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (TST)
Description: The treatment effect of Circadin® 2/5 mg minitabs was compared to that of a placebo on total sleep time, as assessed by the Sleep and Nap Diary questionnaire, following 13 weeks of double-blind treatment
Time Frame: 13 weeks
Population: All patients in the Safety Analysis Set who satisfied all major entry criteria (I.Criteria 1-5) and who had a valid mean TST result recorded for baseline and at least one post-baseline period assessment during the double-blind phase.
  Patients were classified according to randomized treatment. This analysis set was used for all efficacy analyses.
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- Circadin 2/5/10 mg: Circadin 2/5/10 mg: Active arm Units: minutes arithmetic mean (standard error): 51.03 (±10.46)
- Placebo: Placebo arm Units: minutes arithmetic mean (standard error): 18.71 (±10.82)
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
minutes | 51.03 [30.3 to 71.76] | 18.71 [-2.73 to 40.15]
Statistical Analysis 1: Comparison: Circadin 2/5/10 mg vs Placebo; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Final Values) = 32.32, 95% CI 2-sided [2.38 to 62.26], Standard Error of Mean 15.1

2. Secondary Outcome: Sleep Latency (Mins)
Description: Sleep Latency (minutes) derived from Sleep and Nap Diary following 13 weeks of double-blind treatment with Circadin 2/5 mg minitabs versus placebo.
  The lower the value for sleep latency, the better the outcome.
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
minutes
  Baseline | 95.16 (59.253) | 98.76 (73.899)
  13 weeks | 60.74 (42.111) | 76.88 (82.589)
Statistical Analysis 1: Comparison: Circadin 2/5/10 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = -25.2, 95% CI 2-sided [-44.61 to -5.8], Standard Error of Mean 9.787

3. Secondary Outcome: Duration of Wake After Sleep
Description: Duration of Wake after Sleep onset period derived from Sleep and Nap Diary following 13 weeks of double-blind treatment with Circadin 2/5 mg minitabs versus placebo.
  The shorter the value, the better the outcome.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
minutes
  Baseline | 64.4 (24.421) | 64.89 (32.525)
  13 weeks | 68.75 (32.199) | 70.89 (51.590)

4. Secondary Outcome: Number of Awakenings Per Night
Description: Number of awakenings per night will be assessed by a Sleep and Nap Diary and summarized after 13 weeks of double-blind treatment for each treatment group using descriptive statistics.
  The smaller the number, the better the outcome.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Number of awakenings per night
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
Number of awakenings per night
  Baseline | 2.11 (1.655) | 1.92 (1.441)
  13 weeks | 2.37 (2.095) | 2.14 (1.895)

5. Secondary Outcome: Longest Sleep Period
Description: The longest sleep period following 13 weeks of double-blind treatment with Circadin 2/5 mg and placebo was evaluated by a Sleep and Nap Diary questionnaire.
  The longer the sleep period, the better the outcome.
Time Frame: 13 weeks
Population: FAS (Full analysis set)
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Placebo: placebo group
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
minutes
  Baseline | 383.79 (117.677) | 380.58 (118.429)
  13 weeks | 451.45 (124.933) | 414.65 (124.993)
Statistical Analysis 1: Comparison: Circadin 2/5/10 mg vs Placebo; Mixed Models for Repeated Measures (MMRM) analysis; Test type: Superiority; p = 0.053, MMRM
Statistical Analysis 2: Comparison: Circadin 2/5/10 mg vs Placebo; Test type: Superiority; p = 0.039, MI analysis

6. Secondary Outcome: Social Functioning - Children Global Assessment Scale (CGAS)
Description: The Children's Global Assessment Scale (CGAS) Questionnaire measures social functioning at home, in school, and in community settings.
  The scores range from 1, which is the very worst, to 100, which is the very best.
Time Frame: 13 weeks
Population: FAS set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 58 | 61
score on a scale | 48.3 (17.93) | 51.5 (18.02)

7. Secondary Outcome: Behavior at Home and in School - Strengths and Difficulties Questionnaire (SDQ)
Description: The Strengths and Difficulties Questionnaire (SDQ) is a brief, 25-item, measure of behavioral and emotional difficulties that can be used to assess behavior at home and in school in children.
  The SDQ consists of 25 items which are divided into 5 subscales: 1) emotional symptoms (5 items); 2) conduct problems (5 items); 3) hyperactivity/inattention (5 items); 4) peer relationship problems (5 items); and 5) prosocial behavior (5 items).
  Subscales 1 to 4 are summed to generate a Total Difficulties Score (that ranges from 0 to 40). Each item on the SDQ is scored on a 3-point ordinal scale with 0 = not true, 1 = somewhat true, and 2 = certainly true, with higher scores indicating larger problems.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Circadin 2/5/10: Circadin 2/5/10. Active arm
- Placebo: Control group
Arm/Group | Circadin 2/5/10 | Placebo
Number analyzed (Participants) | 58 | 61
score on a scale | 19.6 (5.09) | 20.7 (6.09)
Statistical Analysis 1: Comparison: Circadin 2/5/10 vs Placebo; Test type: Superiority; p = 0.077, MMRM

8. Secondary Outcome: Number of Dropouts
Description: Number of dropouts during the 13 weeks of double-blind treatment in the Circadin 2/5 mg and placebo arms.
Time Frame: 13 weeks
Population: Safety set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo. Control group
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 60 | 65
Participants | 9 | 21
Statistical Analysis 1: Comparison: Circadin 2/5/10 mg vs Placebo; Test type: Superiority; p = 0.04, Chi-squared

9. Secondary Outcome: Assessment of Sleep Parameters by Actigraphy
Description: Actigraphy is a validated method of objectively measuring sleep parameters and average motor activity over days to weeks using a noninvasive device.
  Despite major efforts to ensure adherence, actigraphy monitoring was challenging in this population, and a majority of patients (75% in the Circadin and 77% in the placebo group) refused to wear the device and/or took it off sometime during the night. Only 12 patients in the Circadin and 13 in the placebo group had data for both baseline and 13 weeks of treatment, and even in those it was not possible to ascertain that they wore the device throughout the night.
Time Frame: 13 weeks
Population: Despite major efforts to ensure adherence, actigraphy monitoring was challenging in this population, and a majority of patients (75% in the Circadin and 77% in the placebo group) refused to wear the device during one or both periods and/or took it off some time during the night. Only 12 patients in the Circadin and 13 in the placebo group had data for both baseline and 13 weeks of treatment, and even in those it was not possible to ascertain that they wore the device throughout the night.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 12 | 13
minutes
  Change in TST (total sleep time) | 7.23 (96.521) | -23.94 (61.860)
  Change in sleep latency | 25.11 (38.371) | -12.50 (24.744)

10. Secondary Outcome: Safety and Tolerability - Treatment Emergent Signs and Symptoms (TESS) Summary.
Description: Treatment Emergent Signs and Symptoms (TESS). Signs and symptoms not seen at baseline (i.e. before starting the treatment) and/or worsened even if present at baseline.
Time Frame: 13 weeks, 26 weeks, 52 weeks.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 60 | 65
Participants
  Somnolence - Baseline: No Symptoms | 33 | 41
  Somnolence - Baseline: Mild | 10 | 11
  Somnolence - Baseline: Moderate | 13 | 11
  Somnolence - Baseline: Severe | 4 | 2
  Somnolence - 13 weeks: No Symptoms | 42 | 53
  Somnolence - 13 weeks: Mild | 8 | 11
  Somnolence - 13 weeks: Moderate | 6 | 0
  Somnolence - 13 weeks: Severe | 4 | 1
  Somnolence - 26 weeks: No Symptoms | 45 | 51
  Somnolence - 26 weeks: Mild | 4 | 13
  Somnolence - 26 weeks: Moderate | 9 | 1
  Somnolence - 26 weeks: Severe | 2 | 0
  Somnolence - 52 weeks: No Symptoms | 47 | 56
  Somnolence - 52 weeks: Mild | 9 | 9
  Somnolence - 52 weeks: Moderate | 4 | 0
  Somnolence - 52 weeks: Severe | 0 | 0
  Fatigue - Baseline: No Symptoms | 30 | 32
  Fatigue - Baseline: Mild | 13 | 15
  Fatigue - Baseline: Moderate | 11 | 10
  Fatigue - Baseline: Severe | 6 | 8
  Fatigue - 13 weeks: No Symptoms | 33 | 47
  Fatigue - 13 weeks: Mild | 16 | 12
  Fatigue - 13 weeks: Moderate | 9 | 4
  Fatigue - 13 weeks: Severe | 2 | 2
  Fatigue - 26 weeks: No Symptoms | 39 | 49
  Fatigue - 26 weeks: Mild | 14 | 9
  Fatigue - 26 weeks: Moderate | 6 | 7
  Fatigue - 26 weeks: Severe | 1 | 0
  Fatigue - 52 weeks: No Symptoms | 44 | 52
  Fatigue - 52 weeks: Mild | 13 | 9
  Fatigue - 52 weeks: Moderate | 3 | 4
  Fatigue - 52 weeks: Severe | 0 | 0
  Increased Excitability - Baseline: No Symptoms | 25 | 32
  Increased Excitability - Baseline: Mild | 17 | 8
  Increased Excitability - Baseline: Moderate | 11 | 16
  Increased Excitability - Baseline: Severe | 7 | 9
  Increased Excitability - 13 weeks: No Symptoms | 34 | 42
  Increased Excitability - 13 weeks: Mild | 8 | 8
  Increased Excitability - 13 weeks: Moderate | 10 | 9
  Increased Excitability - 13 weeks: Severe | 8 | 6
  Increased Excitability - 26 weeks: No Symptoms | 35 | 49
  Increased Excitability - 26 weeks: Mild | 6 | 7
  Increased Excitability - 26 weeks: Moderate | 12 | 6
  Increased Excitability - 26 weeks: Severe | 7 | 3
  Increased Excitability - 52 weeks: No Symptoms | 42 | 52
  Increased Excitability - 52 weeks: Mild | 3 | 2
  Increased Excitability - 52 weeks: Moderate | 9 | 10
  Increased Excitability - 52 weeks: Severe | 6 | 1
  Dizziness - Baseline: No Symptoms | 56 | 64
  Dizziness - Baseline: Mild | 3 | 1
  Dizziness - Baseline: Moderate | 1 | 0
  Dizziness - Baseline: Severe | 0 | 0
  Dizziness - 13 weeks: No Symptoms | 57 | 64
  Dizziness - 13 weeks: Mild | 3 | 1
  Dizziness - 13 weeks: Moderate | 0 | 0
  Dizziness - 13 weeks: Severe | 0 | 0
  Dizziness - 26 weeks: No Symptoms | 59 | 65
  Dizziness - 26 weeks: Mild | 0 | 0
  Dizziness - 26 weeks: Moderate | 1 | 0
  Dizziness - 26 weeks: Severe | 0 | 0
  Dizziness - 52 weeks: No Symptoms | 60 | 64
  Dizziness - 52 weeks: Mild | 0 | 1
  Dizziness - 52 weeks: Moderate | 0 | 0
  Dizziness - 52 weeks: Severe | 0 | 0
  Hangover Feelings - Baseline: No Symptoms | 52 | 60
  Hangover Feelings - Baseline: Mild | 8 | 4
  Hangover Feelings - Baseline: Moderate | 0 | 1
  Hangover Feelings - Baseline: Severe | 0 | 0
  Hangover Feelings - 13 weeks: No Symptoms | 52 | 61
  Hangover Feelings - 13 weeks: Mild | 6 | 2
  Hangover Feelings - 13 weeks: Moderate | 2 | 2
  Hangover Feelings - 13 weeks: Severe | 0 | 0
  Hangover Feelings - 26 weeks: No Symptoms | 55 | 64
  Hangover Feelings - 26 weeks: Mild | 3 | 0
  Hangover Feelings - 26 weeks: Moderate | 2 | 1
  Hangover Feelings - 26 weeks: Severe | 0 | 0
  Hangover Feelings - 52 weeks: No Symptoms | 57 | 64
  Hangover Feelings - 52 weeks: Mild | 2 | 1
  Hangover Feelings - 52 weeks: Moderate | 1 | 0
  Hangover Feelings - 52 weeks: Severe | 0 | 0
  Mood Swings - Baseline: No Symptoms | 24 | 33
  Mood Swings - Baseline: Mild | 13 | 10
  Mood Swings - Baseline: Moderate | 21 | 14
  Mood Swings - Baseline: Severe | 2 | 8
  Mood Swings - 13 weeks: No Symptoms | 28 | 41
  Mood Swings - 13 weeks: Mild | 15 | 13
  Mood Swings - 13 weeks: Moderate | 13 | 6
  Mood Swings - 13 weeks: Severe | 4 | 5
  Mood Swings - 26 weeks: No Symptoms | 31 | 45
  Mood Swings - 26 weeks: Mild | 13 | 9
  Mood Swings - 26 weeks: Moderate | 13 | 8
  Mood Swings - 26 weeks: Severe | 3 | 3
  Mood Swings - 52 weeks: No Symptoms | 40 | 50
  Mood Swings - 52 weeks: Mild | 10 | 8
  Mood Swings - 52 weeks: Moderate | 6 | 6
  Mood Swings - 52 weeks: Severe | 4 | 1
  Tremor - Baseline: No Symptoms | 55 | 64
  Tremor - Baseline: Mild | 4 | 1
  Tremor - Baseline: Moderate | 1 | 0
  Tremor - Baseline: Severe | 0 | 0
  Tremor - 13 weeks: No Symptoms | 57 | 63
  Tremor - 13 weeks: Mild | 3 | 1
  Tremor - 13 weeks: Moderate | 0 | 1
  Tremor - 13 weeks: Severe | 0 | 0
  Tremor - 26 weeks: No Symptoms | 58 | 65
  Tremor - 26 weeks: Mild | 0 | 0
  Tremor - 26 weeks: Moderate | 2 | 0
  Tremor - 26 weeks: Severe | 0 | 0
  Tremor - 52 weeks: No Symptoms | 56 | 65
  Tremor - 52 weeks: Mild | 2 | 0
  Tremor - 52 weeks: Moderate | 2 | 0
  Tremor - 52 weeks: Severe | 0 | 0
  Seizures - Baseline: No Symptoms | 60 | 64
  Seizures - Baseline: Mild | 0 | 1
  Seizures - Baseline: Moderate | 0 | 0
  Seizures - Baseline: Severe | 0 | 0
  Seizures - 13 weeks: No Symptoms | 60 | 64
  Seizures - 13 weeks: Mild | 0 | 0
  Seizures - 13 weeks: Moderate | 0 | 1
  Seizures - 13 weeks: Severe | 0 | 0
  Seizures - 26 weeks: No Symptoms | 60 | 63
  Seizures - 26 weeks: Mild | 0 | 2
  Seizures - 26 weeks: Moderate | 0 | 0
  Seizures - 26 weeks: Severe | 0 | 0
  Seizures - 52 weeks: No Symptoms | 59 | 64
  Seizures - 52 weeks: Mild | 0 | 1
  Seizures - 52 weeks: Moderate | 1 | 0
  Seizures - 52 weeks: Severe | 0 | 0
  Headache - Baseline: No Symptoms | 47 | 56
  Headache - Baseline: Mild | 7 | 7
  Headache - Baseline: Moderate | 6 | 2
  Headache - Baseline: Severe | 0 | 0
  Headache - 13 weeks: No Symptoms | 49 | 59
  Headache - 13 weeks: Mild | 9 | 4
  Headache - 13 weeks: Moderate | 2 | 1
  Headache - 13 weeks: Severe | 0 | 1
  Headache - 26 weeks: No Symptoms | 54 | 61
  Headache - 26 weeks: Mild | 5 | 3
  Headache - 26 weeks: Moderate | 1 | 1
  Headache - 26 weeks: Severe | 0 | 0
  Headache - 52 weeks: No Symptoms | 53 | 57
  Headache - 52 weeks: Mild | 6 | 7
  Headache - 52 weeks: Moderate | 1 | 1
  Headache - 52 weeks: Severe | 0 | 0
  Nausea/ Vomiting - Baseline: No Symptoms | 52 | 60
  Nausea/ Vomiting - Baseline: Mild | 6 | 5
  Nausea/ Vomiting - Baseline: Moderate | 2 | 0
  Nausea/ Vomiting - Baseline: Severe | 0 | 0
  Nausea/ Vomiting - 13 weeks: No Symptoms | 49 | 57
  Nausea/ Vomiting - 13 weeks: Mild | 7 | 6
  Nausea/ Vomiting - 13 weeks: Moderate | 4 | 2
  Nausea/ Vomiting - 13 weeks: Severe | 0 | 0
  Nausea/ Vomiting - 26 weeks: No Symptoms | 51 | 61
  Nausea/ Vomiting - 26 weeks: Mild | 8 | 4
  Nausea/ Vomiting - 26 weeks: Moderate | 0 | 0
  Nausea/ Vomiting - 26 weeks: Severe | 1 | 0
  Nausea/ Vomiting - 52 weeks: No Symptoms | 53 | 62
  Nausea/ Vomiting - 52 weeks: Mild | 6 | 3
  Nausea/ Vomiting - 52 weeks: Moderate | 1 | 0
  Nausea/ Vomiting - 52 weeks: Severe | 0 | 0
  Rash - Baseline: No Symptoms | 56 | 58
  Rash - Baseline: Mild | 3 | 5
  Rash - Baseline: Moderate | 1 | 2
  Rash - Baseline: Severe | 0 | 0
  Rash - 13 weeks: No Symptoms | 56 | 61
  Rash - 13 weeks: Mild | 3 | 3
  Rash - 13 weeks: Moderate | 0 | 1
  Rash - 13 weeks: Severe | 1 | 0
  Rash - 26 weeks: No Symptoms | 56 | 60
  Rash - 26 weeks: Mild | 2 | 5
  Rash - 26 weeks: Moderate | 2 | 0
  Rash - 26 weeks: Severe | 0 | 0
  Rash - 52 weeks: No Symptoms | 55 | 62
  Rash - 52 weeks: Mild | 4 | 3
  Rash - 52 weeks: Moderate | 1 | 0
  Rash - 52 weeks: Severe | 0 | 0
  Hypothermia - Baseline: No Symptoms | 56 | 63
  Hypothermia - Baseline: Mild | 2 | 1
  Hypothermia - Baseline: Moderate | 2 | 1
  Hypothermia - Baseline: Severe | 0 | 0
  Hypothermia - 13 weeks: No Symptoms | 57 | 62
  Hypothermia - 13 weeks: Mild | 2 | 2
  Hypothermia - 13 weeks: Moderate | 1 | 1
  Hypothermia - 13 weeks: Severe | 0 | 0
  Hypothermia - 26 weeks: No Symptoms | 58 | 64
  Hypothermia - 26 weeks: Mild | 2 | 1
  Hypothermia - 26 weeks: Moderate | 0 | 0
  Hypothermia - 26 weeks: Severe | 0 | 0
  Hypothermia - 52 weeks: No Symptoms | 59 | 65
  Hypothermia - 52 weeks: Mild | 1 | 0
  Hypothermia - 52 weeks: Moderate | 0 | 0
  Hypothermia - 52 weeks: Severe | 0 | 0
  Coughing/ Breathlessness - Baseline: No Symptoms | 49 | 54
  Coughing/ Breathlessness - Baseline: Mild | 7 | 8
  Coughing/ Breathlessness - Baseline: Moderate | 3 | 2
  Coughing/ Breathlessness - Baseline: Severe | 1 | 1
  Coughing/ Breathlessness - 13 weeks: No Symptoms | 48 | 55
  Coughing/ Breathlessness - 13 weeks: Mild | 10 | 7
  Coughing/ Breathlessness - 13 weeks: Moderate | 1 | 2
  Coughing/ Breathlessness - 13 weeks: Severe | 1 | 1
  Coughing/ Breathlessness - 26 weeks: No Symptoms | 55 | 55
  Coughing/ Breathlessness - 26 weeks: Mild | 4 | 7
  Coughing/ Breathlessness - 26 weeks: Moderate | 1 | 3
  Coughing/ Breathlessness - 26 weeks: Severe | 0 | 0
  Coughing/ Breathlessness - 52 weeks: No Symptoms | 54 | 59
  Coughing/ Breathlessness - 52 weeks: Mild | 4 | 5
  Coughing/ Breathlessness - 52 weeks: Moderate | 2 | 1
  Coughing/ Breathlessness - 52 weeks: Severe | 0 | 0
  Other Adverse Event - Baseline: No Symptoms | 48 | 56
  Other Adverse Event - Baseline: Mild | 8 | 7
  Other Adverse Event - Baseline: Moderate | 3 | 1
  Other Adverse Event - Baseline: Severe | 1 | 1
  Other Adverse Event - 13 weeks: No Symptoms | 35 | 48
  Other Adverse Event - 13 weeks: Mild | 18 | 14
  Other Adverse Event - 13 weeks: Moderate | 7 | 3
  Other Adverse Event - 13 weeks: Severe | 0 | 0
  Other Adverse Event - 26 weeks: No Symptoms | 45 | 39
  Other Adverse Event - 26 weeks: Mild | 11 | 15
  Other Adverse Event - 26 weeks: Moderate | 3 | 7
  Other Adverse Event - 26 weeks: Severe | 1 | 4
  Other Adverse Event - 52 weeks: No Symptoms | 35 | 41
  Other Adverse Event - 52 weeks: Mild | 19 | 15
  Other Adverse Event - 52 weeks: Moderate | 6 | 7
  Other Adverse Event - 52 weeks: Severe | 0 | 2

11. Secondary Outcome: Safety and Tolerability - Blood Pressure (mmHg)
Description: Systolic and Diastolic Blood Pressure (mmHg) A normal blood pressure (BP) level is lower than 140/70 mmHg, meaning systolic BP values lower than 140 mmHg, and diastolic BP values lower than 70 mmHg.
  Values within the normal range mean good safety and tolerability outcomes.
Time Frame: 13 weeks, 26 weeks, 52 weeks.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 60 | 65
mmHg
  Diastolic - Baseline | 64.3 (8.31) | 63.9 (10.11)
  Systolic - Baseline | 104.5 (11.37) | 104.7 (13.94)
  Diastolic - 13 weeks | 65.5 (8.74) | 65.9 (10.73)
  Systolic - 13 weeks | 105.5 (11.34) | 106.5 (12.57)
  Diastolic - 26 weeks | 64.5 (9.65) | 65.1 (10.06)
  Systolic - 26 weeks | 105.3 (12.49) | 107.3 (15.46)
  Diastolic - 52 weeks | 65.8 (7.94) | 66.2 (9.84)
  Systolic - 52 weeks | 106.9 (12.81) | 108.1 (14.46)

12. Secondary Outcome: Safety and Tolerability - Pulse (Beats Per Minute)
Description: Safety and tolerability of Circadin treatment compared to placebo: Pulse rate. The normal pulse for healthy adults ranges from 60 to 100 beats per minute (bpm).
  Values within the normal range mean good safety and tolerability outcomes.
Time Frame: 13 weeks, 26 weeks, 52 weeks.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Circadin 2/5/10 mg | Placebo
Number analyzed (Participants) | 60 | 65
beats per minute
  Baseline | 89.2 (13.84) | 92.3 (21.42)
  13 weeks | 90.7 (15.98) | 94.4 (17.96)
  26 weeks | 86.1 (13.01) | 97 (20.16)
  52 weeks | 86.5 (14.46) | 94.2 (19.14)

13. Secondary Outcome: Safety and Tolerability - Respiratory Rate (Bpm)
Description: Respiratory rate (breaths per minute). The normal respiratory rate for elderly individuals living independently is 12-18 breaths per minute while it is 16-25 breaths per minute for those needing long-term care.
  Values within the normal range mean good safety and tolerability outcomes.
Time Frame: 13 weeks, 26 weeks, 52 weeks.
Population: Safety set
Measure: Mean (Standard Deviation); unit: breaths per minute
Groups:
- Circadin 2/5/10: Circadin 2/5/10 mg: Active arm
Arm/Group | Circadin 2/5/10 | Placebo
Number analyzed (Participants) | 60 | 65
breaths per minute
  Baseline | 19.2 (3.40) | 19.6 (4.33)
  13 weeks | 19.2 (3.38) | 19.4 (4.36)
  26 weeks | 18.7 (3.77) | 20 (4.97)
  52 weeks | 18.4 (3.84) | 18.7 (4.30)

14. Secondary Outcome: Safety and Tolerability - Body Temperature (°C)
Description: Body Temperature (°C). Normal body temperature varies by person, age, activity, and time of day. It ranges from 36.1°C to 37.2°C.
  Values within the normal range mean good safety and tolerability outcomes.
Time Frame: 13 weeks, 26 weeks, 52 weeks.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Circadin 2/5/10 | Placebo
Number analyzed (Participants) | 60 | 65
°C
  Baseline | 36.69 (0.479612) | 36.54 (0.684174)
  13 weeks | 36.68 (0.464637) | 36.63 (0.369984)
  26 weeks | 36.76 (0.459521) | 36.57 (0.371819)
  52 weeks | 36.70 (0.457630) | 36.65 (0.439824)

ADVERSE EVENTS:
Time Frame: 104 weeks
Groups:
- Circadin 2/5/10 mg Double Blind: Circadin 2/5/10 mg. Double blind period, active arm
- Circadin 2/5/10 mg Open Label: Circadin 2/5/10 mg. Open-label period, active arm
Arm/Group | Circadin 2/5/10 mg Double Blind | Placebo | Circadin 2/5/10 mg Open Label
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/65 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/65 | 6/95
Other Adverse Events (participants affected / at risk) | 51/60 | 50/65 | 80/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circadin 2/5/10 mg Double Blind (N=60) | Placebo (N=65) | Circadin 2/5/10 mg Open Label (N=95)
SAE - Serious adverse event (Infections and infestations) | 0 | 1 (1) | 2 (2) — PNEUMONIA EYE INFECTION OTITIS MEDIA ACUTE
SAE -Serious adverse event (Gastrointestinal disorders) | 0 | 0 (0) | 1 (1) — CONSTIPATION
SAE -Serious adverse event (Psychiatric disorders) | 0 | 0 | 3 (3) — AGGRESSION OPPOSITIONAL DEFIANT DISORDER Abnormal behaviour
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circadin 2/5/10 mg Double Blind (N=60) | Placebo (N=65) | Circadin 2/5/10 mg Open Label (N=95)
Non-serious adverse events (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 10 (10) | 37 (50) — COUGH DYSPNOEA ASTHMA RHINORRHOEA
Non-serious adverse events (Nervous system disorders) | 25 (26) | 12 (12) | 42 (51) — SOMNOLENCE HEADACHE
Non-serious adverse events (General disorders) | 23 (28) | 19 (28) | 39 (49) — FATIGUE PYREXIA HANGOVER
Non-serious adverse events (Gastrointestinal disorders) | 15 (15) | 15 (18) | 40 (58) — VOMITING DIARRHOEA NAUSEA CONSTIPATION
Non-serious adverse events (Psychiatric disorders) | 21 (22) | 18 (20) | 36 (47) — MOOD SWINGS AGITATION ANXIETY AGGRESSION
Non-serious adverse events (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 10 (10) — Rash
Non-serious adverse events (Infections and infestations) | 9 (9) | 7 (8) | 46 (61) — UPPER RESPIRATORY TRACT INFECTION INFLUENZA OTITIS MEDIA GASTROENTERITIS NASOPHARYNGITIS SINUSITIS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT01906866/Prot_002.pdf
  • Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT01906866/SAP_003.pdf